CLINICAL TRIAL: NCT06956534
Title: Definition, Assessment and Treatment of Spasticity According to Physiotherapists and Occupational Therapists in Flanders, Belgium: A Cross-sectional Qualitative Study.
Status: Completed | Type: Observational
Sponsor: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Wim Saeys, Professor, PhD, MSc, Universiteit Antwerpen
Other Study IDs: 6901
Record Dates: First submitted 2025-04-24; First posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Spasticity
Keywords: spasticity; questionnaire; occupational therapy; physiotherapy
MeSH Terms: conditions — Muscle Spasticity | interventions — Surveys and Questionnaires; Restraint, Physical

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- caregivers: physiotherapists and occupational therapists
  Interventions: Other: Questionnaire and Physical Exam

INTERVENTIONS:
Other: Questionnaire and Physical Exam — online digital questionnaire

SUMMARY:
The definition of spasticity described by Lance in 1980 provided a strong academic foundation for characterizing this neurological symptom. However, there are doubts about its value in clinical practice for evaluating and treating spasticity. This "upper motor neuron syndrome" is highly complex and does not exist in isolation. Beyond the various definitions that have been attributed to it, spasticity correlates with sensory input, movement, muscle properties, and the continuity of the central nervous system. This has led to an ongoing academic debate regarding how spasticity should be classified and how it should be treated correctly.

This study aims to improve quality by gaining a better understanding of how healthcare providers (physiotherapists & occupational therapists) perceive the definition, evaluation, and treatment of spasticity. The questionnaire is based on the existing study by Blanchette et al. (2017), which was conducted in Canada and surveyed both English- and French-speaking physiotherapists and occupational therapists. That study examined sociodemographic data, work environment, satisfaction with measurement tools for spasticity, and treatment preferences. This study adopts these components while adding an extra item: the definition of spasticity. The research team included this item to explore how healthcare providers interpret spasticity. This will be assessed through multiple-choice and open-ended questions.

The research will be conducted under the supervision of Prof. Dr. Steven Truijen (Universiteitsplein 1, 2610 Wilrijk, Belgium, steven.truijen@uantwerpen.be) and Prof. Dr. Wim Saeys (Universiteitsplein 1, 2610 Wilrijk, Belgium, wim.saeys@uantwerpen.be), organized by the University of Antwerp. During this study, no costs or reimbursements will be expected from participants, health insurance, or the research environment.

DETAILED DESCRIPTION:
The questionnaire will be distributed online using the REDCAP data collection system on social media platform, via mail and Linkedin. Official representative groups (occupational therapists and physiotherapists) will be contacted to distribute the Questionnaire QR-code or link to their members.

Participants will be first asked for their consent and informed this study followed all the European GDPR guidelines.

The included respondent group consisted of Dutch-speaking Belgian adults with a degree in physiotherapy or occupational therapy, who completed the full online questionnaire on spasticity. Respondents who did not meet these criteria or who did not confirm the informed consent, were excluded. Experience in the work field was not a requirement to participate in this study. The researchers chose to only include fully completed questionnaires, even if a partially completed questionnaire had some relevant information to process. This was done to be consistent in the number of responses and the data analysis. It is also not known why a respondent chose to stop without filling out all the questions.

In Belgium, occupational therapy is offered as a three-year bachelor's program. Physical therapy, which was originally a three-year bachelor's degree as well, became an academic program of four years in 1998 and was subsequently extended to a five-year master's program in 2002.

Recruitment was carried out by sharing the questionnaires URL link and QR-code on social media and with professional associations for PTs and OTs in Flanders (Axxon and ergotherapie-belgium.be). Additionally, the questionnaire was distributed by email to personal contacts of the researchers, all of whom hold qualifications in physiotherapy or occupational therapy.

To ensure anonymity, each respondent was assigned a chronological identification number, which made it impossible to identify the respondents from the data collected. The data was only processed by the researchers for the purpose of answering the research question in this study. Participation was completely voluntary, and respondents could terminate filling out the questionnaire at any moment without consequences for them. Respondents did not receive a personal benefit for completing the questionnaire. Respondents were also not automatically notified of the results from this study.

Questionnaire and outcome variables The questionnaire was made through 'Research Electronic Data Capture Platform' (REDCAP), which is a secure, online software platform that is in accordance with the General Data Protection Regulation (GDPR). Before filling out the questionnaire, respondents had to provide informed consent.

The questionnaire is based on the work of Blanchette et al. (2017) and consisted of five sections. Because respondents consisted of PTs and OTs in Flanders, which is the Dutch speaking part of Belgium, the questionnaire was created in Dutch. But since this study will be compiled in English, all questions and answers were translated (attachment 1, table 5).

The first section consists of eight questions on the sociodemographic characteristics of the respondents: profession, gender, age (open-ended question), years of experience in the work field, percentage of neurological patients (NPs) in the respondent's clientele, work environment, specialization and highest level of education. For work environment and specialization there was an 'others' option. If there was no appropriate option listed for that respondent, they could fill this in themselves through an open-ended question. These variables were used to categorize respondents into different groups for further analysis.

The second section is about the interpretation and definition of spasticity and was added compared to the questionnaire of Blanchette et al. (2017). First, respondents were asked to describe spasticity in an open-ended question. To mitigate potential bias in responses to the open-ended question, respondents were required to complete this question before gaining access to the multiple-choice question. This consisted of five definitions - originally formulated by Lance (1980), Young (1994), Pandyan et al. (2005), Dressler et al. (2018) and Li et al. (2021) - or 'none of the above', where they had to indicate which one they preferred.

The evaluation of spasticity was questioned through multiple-choice questions in the third section. First, four multiple-choice questions were shown, namely: 'Who is responsible for the evaluation of spasticity?', 'When does it need to take place?', 'How important is the use of validated and reliable assessment methods?', and 'Which assessment methods do you use to evaluate spasticity?'. For the first and fourth answer there was also an option for 'others' if the respondent wanted to add something. For the fourth question, indicating multiple answers was possible. Next, there was a question about how satisfied the respondent is with six listed measurement tools (range of motion (ROM), clonus, modified Ashworth scale (MAS), modified Tardieu scale (MTS), deep tendon reflexes, functional scales). For each tool they could choose between 'not at all satisfied', 'not satisfied', 'satisfied' or 'very satisfied'.

Finally, there was a section consisting of one multiple-choice question regarding the preferred treatment of spasticity. Here, indicating multiple options was also accepted and 'others' was also possible. However, this section was not shown if the respondent indicated that they do not work with NPs.

Questions are as followed:

Therapist Questionnaire Therapist Sociodemographic Characteristics

1. Profession

   * Occupational Therapist
   * Physiotherapist
   * Trained in both professions
2. Gender

   * Male
   * Female
   * Unknown
3. Age

   __________________________________
4. How many years of experience do you have in clinical practice overall?

   * Less than 1 year
   * Approximately 1 to 3 years
   * Between 4 and 10 years
   * More than 10 years
5. What percentage of your clientele consists of neurological patients?

   * None
   * Less than 30% Therapist Questionnaire
   * 31% - 75%
   * More than 75%
6. How would you best describe your work environment? (multiple answers possible)

   * Hospital
   * Rehabilitation center
   * Institute
   * Private practice
   * Medical-pedagogical institute for children
   * Mental health institute
   * School
   * University
   * University college
   * Home care
   * Other: _____________________________
7. What is your current field of work? (multiple answers possible)

   * Neurology
   * Orthopedics
   * Pediatrics
   * Pulmonology
   * Physical Activity
   * Sports
   * Geriatrics Therapist Questionnaire
   * Psychiatry
8. Highest level of professional education

   * Master's degree
   * Bachelor's degree
9. What is your area of specialization?

   * Neurology
   * Orthopedics/Sports
   * Pediatrics
   * Geriatrics
   * Physical Activity
   * Other: _____________________________ Interpretation and Definition of Spasticity
10. How would you describe spasticity?

    __________________________________________
11. Which of the following definitions of spasticity seems most appropriate to you?

    * [ ] Spasticity is a motor disorder characterized by a velocity-dependent increase in tonic stretch reflexes...
    * [ ] A motor disorder due to abnormal intraspinal processing of primary afferent input.
    * [ ] Impaired sensorimotor control from an upper motor neuron lesion causing involuntary muscle activation.
    * [ ] Involuntary muscle hyperactivity in the presence of central paresis, including various components.

    Therapist Questionnaire
    * [ ] A speed- and length-dependent increase in resistance due to hyperexcitable pathways.
    * [ ] None of the above Evaluation of Spasticity
12. Which healthcare provider should be responsible for evaluating spasticity?

    * Physician
    * Physiotherapist
    * Occupational Therapist
    * Nurse
    * Other: _____________________________
13. When should the evaluation/testing take place?

    * At intake
    * After 3 weeks
    * At hospital discharge (returning home)
    * Periodically
    * During rehabilitation
14. How important is it to use validated and reliable measurement tools for spasticity?

    * Very important
    * Important
    * Neutral
    * Unimportant Therapist Questionnaire
    * Not important at all
15. Which of the following measurement tools do you use to evaluate spasticity?

    * Range of Motion
    * Modified Ashworth Scale
    * Deep Tendon Reflexes
    * Functional Scales
    * Ashworth Scale
    * Torque Measurements
    * Modified Tardieu Scale
    * Clinical Score of Tone
    * Spasm Frequency Scale
    * Composite Spasticity Index
    * Clonus Scale
    * Pendulum Test
    * EMG
    * Other: _____________________________
16. How satisfied are you with the following measurement tools?

    * Tool | Not at all | Not satisfied | Satisfied | Very satisfied |
    * Range of Motion | [ ] | [ ] | [ ] | [ ] |
    * Clonus | [ ] | [ ] | [ ] | [ ] |
    * Modified Ashworth Scale | [ ] | [ ] | [ ] | [ ] | Therapist Questionnaire
    * Modified Tardieu Scale | [ ] | [ ] | [ ] | [ ] |
    * Deep Tendon Reflex | [ ] | [ ] | [ ] | [ ] |
    * Functional Scales | [ ] | [ ] | [ ] | [ ] | Treatment of Spasticity
17. How do you currently treat spasticity?

    * Long-term stretching
    * Long-term ice application
    * Sensory-level stimulation (TENS)
    * Motor-level stimulation
    * Vibration
    * Splinting
    * Positioning
    * Traction
    * Other: _____________________________

ELIGIBILITY:
Inclusion Criteria:

* Licensed Occupational Therapists or Physiotherapists
* Dutch Speaking
* Working in Flanders

Exclusion Criteria:

* Questionnaire not completed
* Informed Consent not given

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The included respondent group consisted of Dutch-speaking Belgian adults with a degree in physiotherapy or occupational therapy, who completed the full online questionnaire on spasticity. Respondents who did not meet these criteria or who did not confirm the informed consent, were excluded. Experience in the work field was not a requirement to participate in this study. The researchers chose to only include fully completed questionnaires, even if a partially completed questionnaire had some relevant information to process. This was done to be consistent in the number of responses and the data analysis. It is also not known why a respondent chose to stop without filling out all the questions.
  In Belgium, occupational therapy is offered as a three-year bachelor's program. Physical therapy, which was originally a three-year bachelor's degree as well, became an academic program of four years in 1998 and was subsequently extended to a five-year master's program in 2002.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2024-09-16 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Demographics of professional (Occupational therapists & Physiotherapists) | Once in questionnaire
  1. Profession
     * Occupational Therapist
     * Physiotherapist
     * Trained in both professions
  2. Gender
     * Male
     * Female
     * Unknown
  3. Age
  4. How many years of experience do you have in clinical practice overall?
     * Less than 1 year
     * Approximately 1 to 3 years
     * Between 4 and 10 years
     * More than 10 years
  5. What percentage of your clientele consists of neurological patients?
     * None
     * Less than 30%
     * 31% - 75%
     * More than 75%
  6. How would you best describe your work environment? (multiple answers possible)
     * Hospital
     * Rehabilitation center
     * Institute
     * Private practice
     * Medical-pedagogical institute for children
     * Mental health institute
     * School
     * University
     * University college
     * Home care
     * Other:
  7. What is your current field of work? (multiple answers possible)
     * Neurology
     * Orthopedics
     * Pediatrics
     * Pulmonology
     * Physical Activity
     * Sports
     * Geriatrics
     * Psychiatry
  8. High level of professional education
     * Master's degree
     * Bachelor's degree
  9. What is your area of specialization?
Interpretation and Definition of Spasticity | Once in questionnaire
  10. How would you describe spasticity?
  __________________________________________ 11. Which of the following definitions of spasticity seems most appropriate to you?
  * [ ] Spasticity is a motor disorder characterized by a velocity-dependent increase in tonic stretch reflexes...
  * [ ] A motor disorder due to abnormal intraspinal processing of primary afferent input.
  * [ ] Impaired sensorimotor control from an upper motor neuron lesion causing involuntary muscle activation.
  * [ ] Involuntary muscle hyperactivity in the presence of central paresis, including various components.
  * [ ] A speed- and length-dependent increase in resistance due to hyperexcitable pathways.
  * [ ] None of the above
Spasticity Assessment | Once in questionnaire
  12. Which healthcare provider should be responsible for evaluating spasticity?
  * Physician
  * Physiotherapist
  * Occupational Therapist
  * Nurse
  * Other:
    13. When should the evaluation/testing take place?
  * At intake
  * After 3 weeks
  * At hospital discharge (returning home)
  * Periodically
  * During rehabilitation 14. How important is it to use validated and reliable measurement tools for spasticity?
  * Very important
  * Important
  * Neutral
  * Unimportant Therapist Questionnaire
  * Not important at all 15. Which of the following measurement tools do you use to evaluate spasticity?
  * Range of Motion
  * Modified Ashworth Scale Deep Tendon Reflexes
  * Functional Scales
  * Ashworth Scale
  * Torque Measurements
  * Modified Tardieu Scale
  * Clinical Score of Tone
  * Spasm Frequency Scale
  * Composite Spasticity Index
  * Clonus Scale
  * Pendulum Test
  * EMG
  * Other:
    16. How satisfied are you with the following measurement tools? Range of Motion Clonus Modified Ashworth Scale Deep Tendon Reflex Functional Scal
Spasticity Management | Once in questionnaire
  17. How do you currently treat spasticity?
  * Long-term stretching
  * Long-term ice application
  * Sensory-level stimulation (TENS)
  * Motor-level stimulation
  * Vibration
  * Splinting
  * Positioning
  * Traction
  * Other: _____________________________

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Rehabilitation sciences and physiotherapy (MOVANT), Antwerp, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Data Available on REDCAP platform. Link and entry approval can be asked to our DPO commisioner
Supporting Information: Study Protocol, CSR
Time Frame: From publication ( around June 2025) and afterwards 20 years (limit of data storage)
Access Criteria: University or Academic Institution